CLINICAL TRIAL: NCT06409338
Title: Research on the Brain Mechanism of Transcutaneous Auricular Vagus Nerve Stimulation in Regulating PD Motor Symptoms
Brief Title: Research on the Brain Mechanism of taVNS in Regulating PD Motor Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-SR-235
Record Dates: First submitted 2024-05-05; First posted 2024-05-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; motor symptoms; taVNS; neural mechanism
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Transcutaneous auricular vagus nerve stimulation (Active Comparator): For Experimental Arm, active transcutaneous auricular vagus nerve stimulation, Patients underwent 14 consecutive daily sessions of taVNS.
  Interventions: Device: Transcutaneous auricular vagus nerve stimulation (active）
- Sham Transcutaneous auricular vagus nerve stimulation (Sham Comparator): For sham transcutaneous auricular vagus nerve stimulation arm, Sham Comparator, patients underwent 14 consecutive daily sessions of sham-taVNS (the electrodes were fixed at the the left earlobe).
  Interventions: Device: Transcutaneous auricular vagus nerve stimulation (sham）

INTERVENTIONS:
Device: Transcutaneous auricular vagus nerve stimulation (active） — Transcutaneous auricular vagus nerve stimulation was conducted by transcutaneous electrical stimulation therapy instrument to the cymba conchae of left ear in the vicinity of the auricular branch vagus nerve. Stimulation parameters: frequency = 20 Hz; pulse width = 500 μs, twice a day, 30 minutes each time.
  Arms: Active Transcutaneous auricular vagus nerve stimulation
Device: Transcutaneous auricular vagus nerve stimulation (sham） — In the sham stimulation group, the electrodes were fixed at the left earlobe with the same stimulus parameters. Stimulation parameters: frequency = 20 Hz; pulse width = 500 μs, twice a day, 30 minutes each time.
  Arms: Sham Transcutaneous auricular vagus nerve stimulation

SUMMARY:
This study is a double blind comparative study exploring the neural underpinnings of taVNS modulating PD motor deficits. We hypothesize that taVNS might improve PD motor deficits by regulating the balance between excitation and inhibition in the primary motor cortex.

DETAILED DESCRIPTION:
Patients in the Experimental group underwent fourteen consecutive daily sessions of transcutaneous auricular vagus nerve stimulation (taVNS, twice daily, 30 minutes each time) , whereas patients in the sham stimulation group underwent fourteen consecutive daily sessions of sham taVNS with the electrodes were fixed at the left earlobe . Assessments of motor symptoms and cortical activity (using Functional near-infrared spectroscopy and Transcranial magnetic stimulation) were performed two times: at baseline, one day post intervention.

ELIGIBILITY:
Inclusion Criteria:

* (1) had a diagnosis of idiopathic PD according to the Movement Disorder Society Clinical Diagnostic Criteria for PD and ON-medication Hoehn and Yahr (H&Y) stage ≤2,
* (2) had stable pharmacotherapy for PD at least one month prior to the study,
* (3) were aged between 40 and 80,
* (4) signed written informed consent,
* (5) can cooperate with the testing and taVNS treatment.

Exclusion Criteria:

* (1) with cognitive impairment, according to Montreal Cognitive Assessment (MOCA) < 24;
* (2) with severe tremor or levodopa-induced dyskinesia;
* (3) with current intake of anticholinergics or any drugs that could induce cerebral functional change;
* (4) with taVNS contraindications;
* (5) received VNS treatment during the past six month;
* (6) with concomitant severe neurologic, renal, cardiovascular, or hepatic disease.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-05-11 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
alterations in functional topological properties within the cortex of bilateral cerebral hemispheres-Sigma | Assessed at baseline, one day post intervention
  Resting state fNIRS data was preprocessed to obtain the cortical oxyhemoglobin values which indicate the cortical excitability. Based on the established cortical functional network, we calculate three typical global parameters named small-worldness (Sigma) which can valuatable cortical network small world attributes.
alterations in functional topological properties within the cortex of bilateral cerebral hemispheres-global efficiency (Eg) | Assessed at baseline, one day post intervention
  Resting state fNIRS data was preprocessed to obtain the cortical oxyhemoglobin values which indicate the cortical excitability. Based on the established cortical functional network, we calculate three typical global parameters named global efficiency (Eg) which can To evaluate the global efficiency of parallel information transmission in cortical networks.
alterations in functional topological properties within the cortex of bilateral cerebral hemispheres-local efficiency (Eloc) | Assessed at baseline, one day post intervention
  Resting state fNIRS data was preprocessed to obtain the cortical oxyhemoglobin values which indicate the cortical excitability. Based on the established cortical functional network, we calculate typical global parameter named local efficiency (Eloc) which can evaluate functional separation in cortical networks.
alterations in functional topological properties within the cortex of bilateral cerebral hemispheres-nodal efficiency (Ne) | Assessed at baseline, one day post intervention
  Resting state fNIRS data was preprocessed to obtain the cortical oxyhemoglobin values which indicate the cortical excitability. Based on the established cortical functional network, we calculate one nodal parameter named nodal efficiency (Ne) which can evaluate the nodal efficiency of information transmission in cortical networks.
changes in MEPs values | Assessed at baseline, one day post intervention
  Surface electromyography (sEMG) recordings from the abductor pollicis brevis (APB) muscle were obtained to record motor evoked potentials (MEPs), which underwent amplification and filtering (bandwidth 20 Hz to 2000 Hz).
changes in RMT values | Assessed at baseline, one day post intervention
  The individual resting motor threshold (RMT) was established as the minimum stimulus intensity required to evoke a MEP peak-to-peak amplitude of at least 0.05 mV in five of ten consecutive trials in a resting muscle.
changes in CSP values | Assessed at baseline, one day post intervention
  The cortical silent period (CSP) was measured by sEMG of the APB following a single TMS pulse at 130% of the RMT to the opposite PMC-UL, while participants were requested to maintain active contraction of the APB at 20% of the maximum force.
changes in SICI values | Assessed at baseline, one day post intervention
  Test stimulus intensity was set according to an unconditioned MEP with an amplitude of ~1 mV. For the conditioning stimulus of SICI and ICF, 80% of RMT was used. We tested interstimulus intervals (ISIs) of 2 and 4 ms for SICI. Each ISI was repeated 10 times to calculate the average value.
changes in ICF values | Assessed at baseline, one day post intervention
  Test stimulus intensity was set according to an unconditioned MEP with an amplitude of ~1 mV. For the conditioning stimulus of SICI and ICF, 80% of RMT was used. We tested interstimulus intervals (ISIs) of 10 and 15 ms for ICF. Each ISI was repeated 10 times to calculate the average value.

SECONDARY OUTCOMES:
Change from Baseline Unified Parkinson's Disease Rating Scale-III at one day post intervention | Assessed at baseline, one day post intervention
  The measure mainly reflects the overall severity of Parkinson's disease motor symptoms. UPDRS III is a motor examination score that includes 14 items such as facial expression, tremor, rigidity, motor delay, posture disorders, and gait examination, with a total score of 0-56 points. The higher the score, the more severe the physical movement symptoms are.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Kezhong, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No